CLINICAL TRIAL: NCT04000451
Title: A Therapy for Improving Symptoms in Patients With Acute Exacerbations of Copd by an Hydrogen-Oxygen Generator With Neburlizer: A Multi-centric, Randomized, Parallel-control and Double-blinded Clinic Study
Brief Title: A Therapy for Improving Symptoms in Patients With Acute Exacerbations of COPD by Hydrogen-Oxygen Generator With Neburlizer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Asclepius Meditec Inc. (Industry)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); The First Hospital of Hebei Medical University (Other); Fudan University (Other); Shanghai Zhongshan Hospital (Other); Shanghai 10th People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Second Hospital of Shanxi Medical University (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Tianjin Medical University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM20180607
Record Dates: First submitted 2019-06-18; First posted 2019-06-27 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Copd Exacerbation Acute
Keywords: Copd Exacerbation Acute; oxygen; oxyhydrogen
MeSH Terms: interventions — Oxygen Inhalation Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxyhydrogen (Experimental): conventional treatment (bronchodilator (LABA,LAMA) with or without ICS)+ hydrogen/ oxygen inhaled
  Interventions: Device: oxyhydrogen; Drug: Conventional treatment
- oxygen (Experimental): conventional treatment (bronchodilator (LABA,LAMA) with or without ICS)+ oxygen inhaled
  Interventions: Device: Oxygen; Drug: Conventional treatment

INTERVENTIONS:
Device: oxyhydrogen — Hydrogen/oxygen mixed gas inhaled(proportion 2:1),3 L/min . 1 hour each time,twice a day(BID).Test Duration is seven days
  Arms: oxyhydrogen
Device: Oxygen — oxygen inhaled,3 L/min . 1 hour each time,twice a day(BID).Test Duration is seven days
  Arms: oxygen
Drug: Conventional treatment — Bronchodilator (LABA,LAMA) with or without ICS.Conventional treatment is invariable with which was given to COPD patients in seven days before the study

SUMMARY:
The purpose for this study is to determine safety and effectiveness of the oxyhydrogen generator with nebulizer through a therapy for improving symptoms in patients with acute exacerbations of copd.

DETAILED DESCRIPTION:
In this study, patients with acute exacerbations of copd who were included in both treatment and control groups, administered randomly oxyhydrogen generator with nebulizer (treatment group) or oxygen Nebulizer Machine (control group for the therapy. The therapeutic outcomes in both treatment and control groups are analyzed and evaluated to verify safety and effectiveness of the test product. This study is a multi-center, randomized, double-blind study. The trial lasted for about 10 days. The curative effect was observed for subjects in the First, the second, the third, the fourth, the fifth, the sixth, the seventh day, respectively as the observing time point. Total patients which are planned to be included are 108 cases, where, 54 cases in the treatment group and control group respectively are distributed in 10 clinical hospitals

ELIGIBILITY:
Inclusion Criteria:

1. meet the diagnostic criteria of chronic obstructive pulmonary disease (COPD)[1] : In the examination of pulmonary function, after inhalation of bronchodilator, the volume of forced air in one second accounted for 70% of forced vital capacity (FEV1 / FVC%) , fev180% ;
2. meet the diagnostic criteria of acute exacerbation of chronic obstructive pulmonary disease (AECOPD)[2] : compared with the stable phase, the patient's condition has continued to deteriorate, more than the normal changes in the daytime, that is, patients with chronic obstructive pulmonary disease foundation for acute onset, need to adjust the routine medication. There are at least 2 of the following 3 items in the continuous deterioration of clinical symptoms: 1 aggravation of shortness of breath; 2 increase of Sputum Volume; 3 purulent sputum; or at least 1 of the above 3 symptoms, but one of the other 5 indicators should be added, 1 fever; 2 increased respiratory frequency and heart rate by 20% compared with the baseline; 3 aggravated cough; 4 Pharyngodynia and runny in the last 5 days; 5 increased wheezing;
3. the age is over 40 years old and has the normal independent judgment ability patient, the male and the female are not limited;
4. AECOPD patients requiring in-patient Care;
5. patients with BCSS score ≥6 at the time of admission;
6. patients who volunteer for the trial and sign an informed consent form.

Exclusion Criteria:

1. screening period of intravenous or oral administration of more than 80 mg / day of methylprednisolone or equivalent dose of other hormones or serious need for continuous non-invasive ventilation patients;
2. having a significant disease other than COPD, which, according to the researchers'judgement, would put the participants at risk for participating in the study or have an impact on the results of the study and the participants'ability to participate in the study;
3. other respiratory diseases: subjects with other active pulmonary diseases, such as active tuberculosis, lung cancer, bronchiectasis disease (CT showed repeated acute exacerbations of bronchiectasis disease) , sarcoidosis, idiopathic interstitial pulmonary fibrosis (IPF) , primary pulmonary hypertension, uncontrolled Sleep apnea (i.e. , according to the researchers, the severity of the disease would influence the study) ;
4. Lung Rehabilitation: Participants in the Lung Rehabilitation Program during the study period;
5. a history of severe heart disease such as acute myocardial infarction, congestive heart failure (NYHA Class III and above) , Severe Arrhythmia and other acute heart disease;
6. serious primary diseases of important organs and systems, such as acute stroke, hypertension above moderate after treatment, active gastric ulcer, diabetes Mellitus (serious complication) , malignant tumor, etc.
7. confirmed and suspected cases of lung cancer;
8. a history of one or more lobectomies;
9. limited understanding and poor compliance;
10. lack of or restricted legal capacity;
11. those who have participated in clinical trials of other drugs or medical devices within 30 days prior to screening but have not reached the end point of the trial;
12. pregnant, lactating women and women of childbearing age who do not agree to effective contraceptive measures during the study period;
13. Persons with mental or physical disabilities;
14. a suspected or confirmed history of alcohol or Drug Abuse;
15. those who are known to be intolerant to inhalation therapy;
16. AST, ALT were 3 times higher than the normal upper limit, creatinine ≥176.8 MMOL / l;
17. shock or other Hemodynamics instability;
18. people with active Hepatitis A, hepatitis B, HIV, tuberculosis, and Infectious Disease Connective Tissue Disease;
19. intravenous hormone therapy for more than 5 days after an acute episode;
20. non expectorant antioxidants, including high doses of vitamin C and Vitamin E;
21. the researcher did not consider it appropriate to participate in this study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
The Breathlessness, Cough, and Sputum Scale(BCSS score) | everyday from the baseline to the seventh day
  The breathlessness, cough and sputum scale (BCSS) is a three-item questionnaire rating breathlessness, cough and sputum on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms).the total total is 12. Variables to be measured or calculated are: from the Baseline to the seventh day.

SECONDARY OUTCOMES:
COPD assessment test (CAT) | baseline and the seventh day
  CAT includes eight items describing the presence or absence of cough, mucus production, chest tightness,ff ort dyspnoea, limitation of activities at home, sense of confidence about leaving the home, sleep and the feeling of having lots of energy. Th e symptoms are assessed on a six-point scale from 0 to 5. Th e main outcome measure is the total score, where 0 indicates the absence of any negative infl uence of disease and 40 the worst imagin-able health status ， Variables to be measured or calculated are: from the Baseline to the seventh day.
FEV1 | baseline and the seventh day
  Change from Baseline in First second forcibly expiration quantity(FEV1) at 7 days
FVC | baseline and the seventh day
  Change from Baseline in Forcibly vital capacity(FVC) at 7 days
FEV1/FVC | baseline and the seventh day
  Change from Baseline in Forced Expiratory Volume in the first second/Forcibly vital capacity(FEV1/FVC) at 7 days
PaO2 | baseline and the seventh day
  Change from Baseline in Arterial oxygen tension (PaO2) at 7 days
PaCO2 | baseline and the seventh day
  Change from Baseline in carbon dioxide arterial tension (PaCO2) at 7 days
Potential of Hydrogen | baseline and the seventh day
  Change from Baseline in Potential of Hydrogen( Ph ) at 7 days
oxygen saturation of blood | everyday from the baseline to the seventh day
  Change from Baseline in oxygen saturation of blood at 7 days
Results Of Performance Evaluation Of Apparatus | everyday from the baseline to the seventh day
  During the treatment period of each subject, the performance of the test instrument must be evaluated from the following 3 aspects every day after treatment, and the percentage of "good" should be calculated.
  Good: The clinical use of the product is more convenient, easy to operate, no fault; General: Normal clinical use of the product, General Operation Requirements, there are occasional small failures.
  Poor: The product is difficult to use, more difficult operation, there are more failures.
  Variables to be measured or calculated are:Results of instrument performance evaluation at the end of each treatment day.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
the main evaluation index and the secondary evaluation index of all participants will be share in 3 months after the end of this study.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Leidy NK, Schmier JK, Jones MK, Lloyd J, Rocchiccioli K. Evaluating symptoms in chronic obstructive pulmonary disease: validation of the Breathlessness, Cough and Sputum Scale. Respir Med. 2003 Jan;97 Suppl A:S59-70. PMID 12564612
- [Background] Leidy NK, Rennard SI, Schmier J, Jones MK, Goldman M. The breathlessness, cough, and sputum scale: the development of empirically based guidelines for interpretation. Chest. 2003 Dec;124(6):2182-91. doi: 10.1378/chest.124.6.2182. PMID 14665499
- [Derived] Zheng ZG, Sun WZ, Hu JY, Jie ZJ, Xu JF, Cao J, Song YL, Wang CH, Wang J, Zhao H, Guo ZL, Zhong NS. Hydrogen/oxygen therapy for the treatment of an acute exacerbation of chronic obstructive pulmonary disease: results of a multicenter, randomized, double-blind, parallel-group controlled trial. Respir Res. 2021 May 13;22(1):149. doi: 10.1186/s12931-021-01740-w. PMID 33985501